CLINICAL TRIAL: NCT05510856
Title: Comparative Clinical Study Evaluating the Possible Efficacy of Duloxetine, Gabapentin and Lacosamide on Oxaliplatin-Induced Peripheral Neuropathy in Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sally Said Mohamed Tantawy, Clinical Pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: oxaliplatin induced neuropathy
Record Dates: First submitted 2022-08-13; First posted 2022-08-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Oncology
Keywords: oxaliplatin,peripheral neuropathy
MeSH Terms: conditions — Neoplasms; Peripheral Nervous System Diseases | interventions — Duloxetine Hydrochloride; Gabapentin; Lacosamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Duloxetine (Experimental): group 1
  Interventions: Other: Duloxetine
- Gabapentin (Experimental): group 2
  Interventions: Other: Gabapentin
- Lacosamide (Experimental): group 3
  Interventions: Other: Lacosamide

INTERVENTIONS:
Other: Duloxetine — Duloxetine 30mg / day for 12 cycles (up to 6 months)
  Arms: Duloxetine
Other: Gabapentin — Gabapentin 300 mg / day for 12 cycles (up to 6 months)
  Arms: Gabapentin
Other: Lacosamide — Lacosamide 50 mg / day for 12 cycles (up to 6 months)
  Arms: Lacosamide

SUMMARY:
This study aims to investigate the possible efficacy of duloxetine, gabapentin and lacosamide on oxaliplatin-induced peripheral neuropathy in patients with gastrointestinal cancer.

DETAILED DESCRIPTION:
This is a randomized, double-blind,controlled, parallel study that will be conducted on patients with oxaliplatin induced peripheral neuropathy with gastrointestinal cancer.

This study will be done on 93 patients with gastrointestinal cancer (colon or gastric or pancreatic) cancer on standard FOLFOX-4 regimen who will divided into 3 groups:

Group 1: 31 Patients who will receive standard chemotherapy plus duloxetine 30 mg/day for 12 cycles (up to 6 months).

Group 2: 31 Patients who will receive standard chemotherapy plus gabapentin 300 mg/day for 12 cycles (up to 6 months).

Group 3: 31 Patients who will receive standard chemotherapy plus lacosamide 50 mg/day for 12 cycles (up to 6 months).

ELIGIBILITY:
Inclusion Criteria:

* A) Adults ≥ 18 years old male and female patients. B) Patients with gastrointestinal cancer receiving oxaliplatin chemotherapy

Exclusion Criteria:

* A) Preexisting neuropathic or brain disorders. B) Previous use of chemotherapeutic agents including taxanes, platinum, vinca alkaloids, and bortezomib.

C) Concomitant use of drugs reported to have neuroprotective role and analgesics.

D) Patients with diabetes, uncontrolled hypertension, congestive heart failure, drug addiction and patients who were receiving tamoxifen.

E) Patients with abnormal renal function tests (serum creatinine ≤ 30 ml/min) or liver function tests (≥ 3 times the upper normal range).

F) Participants with a documented medical history of neuropathy. G) Concomitant use of other antidepressants, anticonvulsants, high-dose vitamin supplements or drugs known to influence serotonin levels.

H) Pregnancy and lactating women. I) Uncooperative patients and patients who have psychological problems or on antipsychotic medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
McGill Pain Questionnaire | every 2 weeks
  questionnaire
12-item neurotoxicity questionnaire | every 4 weeks
  questionnaire
EORTC Core Quality of Life questionnaire | up to 6 months
  questionnaire
Common Terminology Criteria for Adverse Events | every 4 weeks
  questionnaire

SECONDARY OUTCOMES:
Neurofilament light chain (NfL) | up to 6 months
  biological biomarker
Nuclear factor- kappa B (NF- κB) | up to 6 months
  biological biomarker
Neurotensin (NT) | up to 6 months
  biological biomarker
Hemeoxygenase-1 | up to 6 months
  biological biomarker

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Department, Tanta University, Tanta, Egypt